CLINICAL TRIAL: NCT02510339
Title: The Incidence of Associated Intra-articular Knee Pathology With Concomitant Tibial Shaft Fractures Treated With Suprapatellar Nailing
Brief Title: Tibial Shaft Nailing Treated With Suprapatellar Nailing
Status: Completed | Type: Observational
Sponsor: Orlando Health, Inc. (Other)
Responsible Party: Principal Investigator, Paula J. Harriott, Clinical Research Coordinator, Orlando Health, Inc.
Other Study IDs: 15.047.04
Record Dates: First submitted 2015-07-08; First posted 2015-07-29 (Estimated); Last update posted 2017-04-10 (Actual); Status verified 2015-10

CONDITIONS: Broken Leg
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observational: The Lysholm Knee score and the SF-36 questionnairs will be given to patients presenting to Orlando Regional Medical Center with open or closed fractures of the tibial shaft during their follow up visits post operativily.
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — Administration of two questionnairs during post operative visits.

SUMMARY:
The goal of this project is to determine the incidence of intra-articular knee pathology following tibial shaft fractures as evaluated by intraoperative knee aspiration and physical exam, and to evaluate for chondral injuries following treatment with a suprapatellar tibial nail via MRI.

DETAILED DESCRIPTION:
Suprapatellar tibial nailing is gaining popularity throughout the orthopedic community for tibial shaft fractures, however the secondary effects of this technique on the articular cartilage of the knee is unknown. Additionally, the incidence of intra-articular knee pathology in the face of tibial shaft fractures has not been described in the orthopedic literature. An undiagnosed cruciate/collateral ligament injury can result in post-traumatic arthritis, as well as a delay in justified ligamentous reconstruction of the knee, causing further injury. Long term sequelae of now commonplace suprapatellar nailing on the patellofemoral joint of the knee have been sparsely elucidated in the literature.

The primary objective is to determine the consequences of suprapatellar tibial nailing on cartilage of the patellofemoral joint.

As a secondary objective, this study will seek to determine the incidence of intra-articular knee pathology following tibial shaft fractures in patients presenting to Orlando Regional Medical Center.

ELIGIBILITY:
Inclusion Criteria:

1. skeletally mature
2. open or closed fractures of the tibial shaft

Exclusion Criteria:

1. concomitant tibial plateau or tibial pilon injuries
2. a knee dislocation
3. skeletally immature
4. those who will undergo standard (infra-patellar) tibial nailing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include skeletally mature patients of Level One Orthopaedics, presenting to Orlando Regional Medical Center with open or closed fractures of the tibial shaft.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2016-01-10 (Actual); Primary Completion 2017-03-01 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
Consequences of suprapatellar tibial nailing | One year
  During follow up visits, subjects will be given the Olerud-Molander questionnaire to complete. The data from that form will be analyzed for each visit.

SECONDARY OUTCOMES:
Incidences of intra-articular knee pathology | One year.
  Post-operative radiographs will be analyzed during each visit per standard of care.
Functional assessment | One year
  The functional assessment/progress of the patient will be noted at each follow up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Tara Roberts, BS, Study Chair — Orlando Health IRB corporate manager